CLINICAL TRIAL: NCT01906957
Title: Cerebral Oxygenation, Cardiac Output,Cognitive Function, and Exercise Training in Patients With Metabolic Syndrome, Coronary Heart Disease and Chronic Heart Failure.
Brief Title: Cognition and Exercise Training
Acronym: COGNEX-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sufficient financial - staff resources
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Mathieu Gayda, P.hD, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COGNEX-2
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome; Coronary Heart Disease; Chronic Heart Failure
MeSH Terms: conditions — Metabolic Syndrome; Coronary Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Elderly healthy subjects (Experimental): Randomization into :
  1. high intensity interval training (HIIT)(n=20)
     or
  2. moderate intensity intensity continuous exercise (n=20)
  Interventions: Other: high intensity interval training (HIIT); Other: moderate intensity continuous exercise training
- Patients with metabolic syndrome (Experimental): Randomization into :
  1. high intensity interval training (HIIT)(n=20)
     or
  2. moderate intensity intensity continuous exercise (n=20)
  Interventions: Other: high intensity interval training (HIIT); Other: moderate intensity continuous exercise training
- coronary patients (Experimental): Randomization into :
  1. high intensity interval training (HIIT)(n=20)
     or
  2. moderate intensity intensity continuous exercise (n=20)
  Interventions: Other: high intensity interval training (HIIT); Other: moderate intensity continuous exercise training
- heart failure patients (Experimental): Randomization into :
  1. high intensity interval training (HIIT)(n=20)
     or
  2. moderate intensity intensity continuous exercise (n=20)
  Interventions: Other: high intensity interval training (HIIT); Other: moderate intensity continuous exercise training

INTERVENTIONS:
Other: high intensity interval training (HIIT) — High-intensity interval exercise (HIIE) session This HIIE session will be based on a previous study conducted in our laboratory that compared physiological, psychological and electrocardiological tolerance of four different single bouts of HIIE in coronary patients (Guiraud et al. 2010). The selected HIIE session represented the best compromise between safety, time spent at a high level of VO2peak and psychological adherence. This HIIE session consists of a 10-min warm-up at 50% of MAP, followed by two sets of 10 min composed of repeated bouts of 15 s at 100% of MAP interspersed by 15 s of passive recovery. Four minutes of passive recovery were allowed between the two sets, as well as a 5-min cool-down after the last 15-s exercise bout. A total duration of 35 minutes will be employed for this session for coronary artery disease patients, and 22 minutes for chronic heart failure patients (Guiraut et al. 2010 b).
Other: moderate intensity continuous exercise training — Moderate Intensity Continuous Exercise (MICE) session This exercise session will be based on the recommendations of the American Heart Association on exercise prescription in cardiac rehabilitation (Balady et al. 2007), suggesting that exercise intensity should lie between 50% and 80% of maximal aerobic power (MAP). We opted for an intensity of 70% of MAP. Duration will be adjusted to match total energy expenditure of the HIIE, according to the previous methodology method (Guiraud et al. 2010 b). A total duration of 28.7 minutes will be employed in healthy elderly patients, coronary artery disease patients and patients with metabolic syndrom; and 16 minutes in chronic heart failure patients.

SUMMARY:
The aim of study is to investigate the impact of two different training modalities (high intensity interval training (HIIT) versus moderate intensity continuous exercise training (MICET) on cognitive performance, cerebral oxygenation, cardiac output and physical fitness in older healthy adults, patients with metabolic syndrome, coronary heart disease and heart failure. The investigators hypothesized that HIIT modality will lead to a larger improvement in physical fitness (i.e. VO2peak), cardiovascular parameters (cardiac output and stroke volume) and cognitive performance at rest and during submaximal exercise. The primary endpoint will be the improvement in cognitive performance.

ELIGIBILITY:
Inclusion criteria:

Elderly healthy subjects : with no MetS and no-documented CHD, both males and females, aged>60 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living.

Patients with metabolic syndrome and no-documented CHD, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. MetS will be defined according to recent updated criteria: presence of at least three of five criteria, namely abdominal obesity (waist circumference cut-off depending on the recently published ethnic-based variations, triglycerides > 1.70 mmol/l, decreased HDL-cholesterol (< 1.0 mmol/l in men and < 1.3 mmol/l in women), systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg, and FPG > 5.6 mmol/l.

CHD patients, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. Moreover, they must have documented CHD (prior myocardial infarction, prior coronary angiography or angioplasty, or documented myocardial ischemia on myocardial scintigraphy).

Patients with documented stable chronic heart failure will be recruited if they show the following inclusion criteria:

* ≥18 years
* Left ventricular ejection fraction (LVEF) <40% (measured within 6 months of their enrolment by MUGA Scan, echo or radiological ventriculography)
* NYHA functional class I-III
* Optimal therapy at stable doses including a beta-blocker and an ACE inhibitor or ARA for at least 6 weeks prior to investigation (unless documented rationale for variation).
* Able to perform an symptom limited exercise test.
* Capacity and willingness to sign the informed consent form.

Exclusion Criteria:

* For healthy elderly subjects:
* age under 60 years
* lack of expressed written consent
* metabolic syndrome
* coronary heart disease
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* chronic atrial fibrillation
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For patients with metabolic syndrome:

* lack of expressed written consent
* coronary heart disease
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* chronic atrial fibrillation
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For patients with CHD

* lack of expressed written consent
* recent acute coronary event (< 3 months)
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* severe non-revascularize coronary disease including left main coronary stenosis
* patient awaiting coronary artery bypass surgery
* chronic atrial fibrillation
* presence of permanent ventricular pacemaker
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For CHF patients:

* Any relative or absolute contraindications to exercise training among patients with stable chronic heart failure according to current recommendations (Working Group on Cardiac Rehabilitation 2001)
* Fixed-rate pacemaker or ICD devices with heart rate limits set lower than the exercise training target heart rate.
* Major cardiovascular event of procedure within the 3 months preceding enrolment in the study.
* Atrial fibrillation
* Heart failure secondary to significant uncorrected primary valvular disease (except for mitral regurgitation secondary to LV dysfunction)
* Heart failure secondary to congenital heart disease or obstructive cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function assessed by standard pen-paper battery test | At baseline and after 3 months
  a) Digit Span (Forward and Backward) (short-term and working memory), b) Digit Symbol Substitution Test (attention & processing speed), c) Trail making test, part A and B (mental flexibility), d) D-KEFS Color-Word Interference Stroop Test (selective attention and inhibition) and e) Rey Auditory Verbal Learning Test (long-term verbal memory).

SECONDARY OUTCOMES:
Maximal aerobic capacity (VO2max) | At baseline and after 3 months
  Gas exchanges will be measured during maximal incremental test. The highest value reached during the exercise phase of the maximal test (ergocycle) will be considered as the VO2max.

OTHER OUTCOMES:
Maximal cardiac output and stroke volume | At baselin and after 3 months
  Maximal cardiac output and stroke volume wil be measured continuously at rest, during exercise and recovery using an impedance cardiography device.
Cerebral hemodynamics with NIRS | At baseline and after 3 months
  Cerebral oxygenation/perfusion will be measured using near-infrared spectroscopy (NIRS) system during maximal exercise and recovery.
Microvascular function at the forearm level (NIRS) | At baseline and after 3 months
  Microvascular function will be assessed using during reactive hyperemia using near-infra red spectroscopy (NIRS) placed on top of the brachio-radialis muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Gayda, Ph.D, Principal Investigator — Montreal Heart Institute
Locations (2):
- Canada (2):
  - Cardiovascular Prevention and Rehabilitation Centre, Montreal Heart Institute, Montreal, Quebec
  - Cardiovascular Prevention and Rehabilitation Centre (EPIC), Montreal Heart Institute, Montreal, Quebec